CLINICAL TRIAL: NCT05974150
Title: Real World Treatment Experience of Patients With Breast, Lung, Ovarian, Multiple Myeloma, or Acute Myelogenous Leukemia (AML) Using Remote Symptom Monitoring
Brief Title: Real World Treatment Experience of Patients With Breast, Lung, Ovarian, Multiple Myeloma, or Acute Myelogenous Leukemia Using Remote Symptom Monitoring
Status: Recruiting | Type: Observational
Sponsor: Carevive Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: OPT-IN Carevive Registry; NCT05974137 (obsolete NCT alias)
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer; Lung Cancer; Multiple Myeloma; Ovarian Cancer; Acute Myelogenous Leukemia
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Multiple Myeloma; Ovarian Neoplasms; Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Web based survey — online weekly survey

SUMMARY:
The goal of this study is to create a data set to add to Carevive's registry from real world clinical and patient reported data collected using an electronic care planning system (CPS) with remote symptom monitoring that is used in routine care for cancer patients on active treatment.

Patients will complete a baseline survey in person using a secured device or remotely using their own electronic device in a location of their choice. Weekly electronic patient reported outcome (PRO) surveys are collected from the patients using the Carevive platform for a minimum of 12 weeks. Patients may continue weekly surveys as long as they are receiving treatment.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be 18 years of age or older.
* Subjects may be any stage and anywhere in the treatment continuum.
* Subject participants must have a diagnosis of a breast, lung, AML, ovarian cancer or multiple myeloma.
* Subjects must be able to complete on-line surveys using a cell phone, tablet, or computer.
* All participants must be able to understand English.

Exclusion Criteria:

* Any patient who cannot understand written or spoken English.
* Any patient without the ability to complete on-line surveys using a cell phone, tablet, or computer.
* Any patient on a treatment clinical trial.
* Any prisoner and/or other vulnerable persons as defined by NIH (45 CFR 46, Subpart B, C and D).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients receiving cancer treatment for breast, lung, GI or multiple myeloma
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-07-19 (Actual); Primary Completion 2025-11-05 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Create Data Set | 1 year
  The goal of this registry is to create a data set from real world clinical and patient reported data collected using an electronic care planning system (CPS) that is used in routine care for cancer patients on active treatment

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Yale Cancer Center, New Haven, Connecticut
  - Northshore University Health System, Evanston, Illinois
  - Univeristy of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke, Durham, North Carolina
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - University Hospitals Seidman Cancer Center, Cleveland, Ohio
  - Tri-County Hematology & Oncology Associates, Inc., Massillon, Ohio

IPD SHARING:
Plan to Share IPD: No